CLINICAL TRIAL: NCT02545478
Title: Early Detection of Inflammatory Biomarkers in Infection
Brief Title: Biomarkers in Infection
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2005P000116
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Infection; Inflammation
Keywords: septic shock; infection; inflammation; pathologic process; biomarkers
MeSH Terms: conditions — Sepsis; Infections; Inflammation; Shock, Septic; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum and plasma, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected Group: subjects with suspected infection
- Non-infected group: subjects without any infection

SUMMARY:
The purpose of this investigation is to evaluate how early biomarkers of infection and inflammation perform in identifying patients at risk for poor outcome in sepsis and septic shock.

DETAILED DESCRIPTION:
The body's immune system and a subsequent inflammatory response are triggered during infection. The detection of an activated immune system, and an indication of the degree of the host response, is helpful to the clinician both in assessing the severity of infection and in patient treatment and management. Currently, the white blood cell count and the differential are the most common laboratory parameters for measuring host response. The sedimentation rate and CRP are also used to detect inflammation. However, these tests are all imperfect predictors, and a test providing a better assessment of immune response would be helpful to the clinician in patient care. Additionally, understanding host response to infection may be helpful in understanding the biology and pathophysiology of sepsis. There are other biomarkers and inflammatory markers that may be found early in the initial presentation of infection such as cytokines (VEGF IL-1,IL-4,IL-6, IL-10, PAF, TNF, lectins iNoS,etc.) and clotting factors (protein C, d-dimer, complements involved in the clotting cascade, CRP, etc) that may provide a means of early detection of systemic inflammation, cell dysfunction, and related conditions. Early identification of patients at risk for systemic inflammatory syndromes, sepsis and septic shock may help direct patients to earlier antibiotic administration and early intervention with goal directed therapy. It may also serve as a tool for risk stratification when components such as age, comorbid illness and infection type are included.

The endothelium and endothelial cell markers are important in sepsis, yet a somewhat under-studied field of research. Additionally, the endothelium is a key regulator of the microcirculation, a place where oxygen diffusion occurs. One focus of this study is to measure endothelial markers (ie VEGF) and other cytokines with the goal of correlating these markers with severity of sepsis. Another focus is to study the response of various components in the blood, including the leukocytes, red cells, the endothelium, as well as cellular components such as the mitochondria. We will specifically look at alterations in thiamine, Vitamin D, CoQ10,l-carnitine and other nutrients as part of (and as related to) the body's response. Recently, a non-invasive method of assessing microvascular circulation by orthogonal polarization spectral (OPS) imagery has become available using a non-invasive technology known as orthogonal polarization spectroscopy. This technique enables direct visualization and quantification of microcirculatory blood flow, and represents an important surrogate outcome to which endothelial cell marker may be correlated. This will involve placing the microscopy probe gently against the sublingual mucosa and collecting a videotape of the circulation lasting about twenty seconds. This process involves minimal (or no) risk - it is akin to taking a temperature and uses no radiation. This videotape will be examined later by a novel software program that quantifies the circulation and used as an important surrogate outcome measure. Additionally, we are going to perform echocardiography to better understand the heart's response to sepsis, and correlated the molecular responses that we find with the changes in the responses by the heart. In addition, we will assess microvascular flow in the skeletal muscle in the forearm using diffuse correlation spectroscopy (DCS). DCS is a novel technique that can be used to measure peripheral tissue perfusion noninvasively and has the potential to provide insight into microcirculatory health and end-organ perfusion. DCS measurement is performed using a small sensor, similar to a pulse oximeter sensor, that attaches to the skin using adhesive. It uses near-infrared light to illuminate the tissue. The change in the transmitted light through the tissue due to the moving red blood cells is characterized to quantify the microvascular flow. DCS is noninvasive, uses no radiation, and involves minimal (or no) risk. DCS measurement will be performed in conjunction with vascular occlusion test (VOT), which involves having a blood pressure cuff placed on the upper arm to cause occlusion and reperfusion of blood flow distally to measure dynamic changes in microvascular flow. We will measure endothelial glycocalyx degradation products (e.g. heparin sulfate, syndecan, etc) in the urine.

This is a multicenter, observational pilot study which aims to evaluate how early biomarkers of infection an inflammation perform in identifying patients at risk for poor outcomes in sepsis and septic shock. The study will utilize a cohort of patients presenting to the ED with suspected infection as well as non-infected control population.

These patients will be compared with a non-infected population.

Enrolled subjects in the infected group will have blood samples and chart review obtained at enrollment, 24, 48 and 72 hours. For the control group, only a single blood draw will be collected at enrollment. Urine may be collected in a convenience sample of patients

Enrolled subjects will also undergo physiologic assessments using echocardiography, Microscan, Non-invasive cardiac output monitor (NICOM), DCS, extremity temperature as well as End-Tidal C02 measurements if a trained researcher is present.

ELIGIBILITY:
Inclusion Criteria for Infected subjects:

* Age 18 years of age or older
* Confirmed or suspected infection

Inclusion Criteria for Control Subjects:

* Age 18 years of age or older
* A non-infectious clinical presentation to include
* Normal white blood cell count ( > 4,000 and/or < 12,000)
* Normothermia ( > 96.5 and/or less 100.4)
* Absence of the following clinical complaints: productive cough, fever, pyuria, rash
* No evidence of acute coronary syndrome

Exclusion Criteria for Control Subjects:

- Suspected infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with suspected infection as well as a non-infected control population.
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2006-04; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
28 day in-hospital mortality | within 28 days after inclusion
  participants will be followed up for 28 days

SECONDARY OUTCOMES:
Organ Dysfunction assessed by Sepsis-related Organ Failure Assessment (SOFA) Score | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Shapiro, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts